CLINICAL TRIAL: NCT02691975
Title: A Phase I/II, Open-Label, Dose-Escalation and -Expansion, Safety, Pharmacokinetics and Efficacy Study of SHR3680 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Safety and Efficacy Study of SHR3680 in Metastatic Castration-Resistant Prostate Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR3680-001
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Hormone Refractory Prostate Cancer; Metastatic Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SHR3680 (Experimental): Tablet
  Interventions: Drug: SHR3680

INTERVENTIONS:
Drug: SHR3680 — SHR3680 is administrated orally, qd, 28 days as one cycle. Patients may continue SHR3680 until disease progression or unacceptable toxicity.

SUMMARY:
This study evaluates the tolerability, safety, pharmacokinetics and efficacy of SHR3680 in patients with metastatic castration-resistant prostate cancer (mCPRC). All participants will receive SHR3680.

DETAILED DESCRIPTION:
Androgenic signaling plays a pivotal role in the development of prostate cancer. Androgen deprivation therapy is the mainstay treatment for this cancer in the metastatic setting, but the disease eventually develops to castration-resistant prostate cancer (CRPC) mainly due to the overexpression of androgen receptors (AR) and continued AR activation.

SHR3680 is a novel strong AR antagonist. By competitively binding to AR, SHR3680 inhibits androgen-mediated translocation of AR to the nucleus, binding of AR to Deoxyribonucleic acid (DNA), and finally the transcription of AR target genes, thus possibly resulting in a specific and strong anti-tumor effect on prostate cancer. Unlike first-generation AR antagonists (e.g. bicalutamide), which undergoes an antagonist-to-agonist switch to stimulate AR in the setting of AR overexpression in CRPC, SHR3680 is a full antagonist of AR and thus it is supposed to be more effective for the treatment of CRPC.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance scale 0 - 1.
* Life expectancy of more than 6 months.
* Histologically or cytologic confirmed prostate adenocarcinoma without neuroendocrine differentiation or small cell features
* Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy
* Evidence of prostate cancer progression by radiographic or PSA criteria
* Radiological evidence of distant metastatic lesions
* Serum testosterone level < 1.7 nmol/L (50 ng/dL) at the screening visit
* Adequate hepatic, renal, heart, and hematologic functions (platelets > 80 × 10e9/L, neutrophil > 1.5 × 10e9/L, Hb >90 g/L,total bilirubin and creatinine within upper limit of normal(ULN), and serum transaminase≤1.5×the ULN).
* Signed and dated informed consent.Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.

Exclusion Criteria:

* Treatment with androgen receptor antagonists, 5-alpha reductase inhibitors, estrogens, or chemotherapy within 4 weeks of enrollment or plans to initiate treatment with any of these drugs during the study
* Prior treatment with enzalutamide, abiraterone, or ketoconazole for prostate cancer
* History of seizure or any conditions that may predispose to seizure
* Concurrent or planned treatment with corticosteroids, medications known to have seizure potential, or herbal products known to decrease PSA levels
* Planned to initiate any other anti-tumor therapies during the study
* Less than 4 weeks from the last clinical trial
* Evidence of brain metastasis or primary tumors
* Clinically significant cardiovascular diseases
* Abuse of alcohol or drugs
* Severe concurrent disease, infection, or bone metastasis that, in the judgment of the investigator, would make the patient inappropriate for enrollment

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 12 weeks
  For Phase 1 portion of study; maximum-tolerated dose (MTD) will be defined as the maximum dose level at which no more than one out of three subjects experience a dose-limiting toxicity (DLT) within the first 12 weeks of multiple dosing
Radiological progression-free survival | 24 months
  For Phase 2 portion of study

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 24 months
  Adverse events are assessed by CTCAE v4.0
The percentage of patients reaching at least a 50% reduction in prostate specific antigen (PSA) as compared to baseline at 12 weeks | 12 weeks
Time to prostate specific antigen (PSA) progression | 24 months
  Prostate specific antigen (PSA) progression is defined by the Prostate Cancer Clinical Trials Working Group (PCWG2) criteria.
Objective response rate | 24 months
Quality of life | 24 months
  Brief Pain Inventory (Short Form), Functional Assessment of Cancer Therapy-Prostate (v4.0)
Peak plasma concentration (Cmax) | 12 weeks
Area under the plasma concentration versus time curve (AUC） | 12 weeks
T1/2 (Half-life) | 12 weeks
  The time required for the plasma concentration of a drug to be reduced by 50%

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, M.D., Principal Investigator — Fudan University
Locations (12):
- China (12):
  - Beijing Hosptial, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Zhenzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin X, Ji D, Gu W, Han W, Luo H, Du C, Zou Q, Sun Z, He C, Zhu S, Chong T, Yao X, Wan B, Yang X, Bai A, Jin C, Zou J, Ye D. Activity and safety of SHR3680, a novel antiandrogen, in patients with metastatic castration-resistant prostate cancer: a phase I/II trial. BMC Med. 2022 Mar 4;20(1):84. doi: 10.1186/s12916-022-02263-x. PMID 35241087